CLINICAL TRIAL: NCT01219309
Title: Omega-3/Omega-6 Fatty Acids for ADHD. A Randomized Placebo-controlled Trial in Children and Adolescents
Brief Title: Omega-3/Omega-6 Fatty Acids for Attention-Deficit/Hyperactivity Disorder (ADHD): A Trial in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Mats Johnson, Department of Child Psychiatry, Göteborg University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ö761-03
Record Dates: First submitted 2010-04-29; First posted 2010-10-13 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-04

CONDITIONS: ADHD; Reading/Writing Disorder
Keywords: Attention-deficit/hyperactivity disorder; Omega 3/6 fatty acids; Developmental coordination disorder; Reading/writing difficulties.
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Skills Disorders | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega 3/6 treatment (Active Comparator)
  Interventions: Dietary Supplement: Omega 3/6 fatty acids
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo (olive oil)

INTERVENTIONS:
Dietary Supplement: Omega 3/6 fatty acids — 3 capsules bid orally
  Other Names: eyeq
  Arms: Omega 3/6 treatment
Dietary Supplement: Placebo (olive oil) — 3 capsules bid orally
  Arms: Placebo

SUMMARY:
Objective: To assess whether supplementation with Omega 3/6 fatty acids (eye q®) was effective in the treatment of ADHD and its diagnostic subtypes and comorbid conditions, in children and adolescents.

Method: Randomized placebo-controlled one-way crossover trial with 75 children and adolescents aged 8-18 years receiving Omega 3/6 or placebo for three months followed by 3 months with Omega 3/6 for all. ADHD symptoms were measured with the investigator-rated ADHD Rating Scale-IV-Parent Version and the Clinical Global Impression (CGI) scale of symptom severity and impairment.

DETAILED DESCRIPTION:
The study design is a randomised, double-blind placebo-controlled trial with a total duration of 6 months. 50-100 children and adolescents, aged 8-18 years, who meet the DSM-IVÔ criteria for Attention-Deficit/Hyperactivity Disorder (ADHD) of any subtype will be given the opportunity to participate. The study comprises 2 study periods.

Study Period I

This is an assessment/evaluation and drug washout phase of up to 1-3 months for those patients taking any medication excluded by the protocol.

Study Period II

Participants will be randomised to 3 months of treatment with a fixed dose of 6 capsules per day of EyeQ, divided in two daily doses, to supply 558 mg EPA, 174 mg DHA and 60 mg GLA daily, or to placebo. Identical capsules containing olive oil will be used as placebo. Randomisation will be organized by Equazen UK Ltd, who will prepare randomisation numbers to be sent out to the investigation centre. At 3 months a one-way treatment crossover of the placebo-group to active treatment will be made so that both patient groups will receive EyeQ for the remaining 3-month period. Compliance will be ascertained through bi-weekly telephone contacts and at each visit. Compliance is defined as taking the prescribed dosage >70% of the days in a visit interval.

Neuropsychiatric assessment:

DSM IV checklist ADHD-Rating Scale IV - Parent:Inv Clinical Global Impression (CGI) scale GAF-scale

FTF teacher questionnaire SNAP-IV teacher questionnaire Brown's ADD teacher scale

Neuropsychological assessment:

WISC-III® or WAIS-III® VMI Digit span Span-board task Qb-test

Brown's ADD self report CDI (Children's Depression Inventory)

Five to Fifteen (FTF) parent questionnaire Brown's ADD parent scale SNAP-IV parent questionnaire Nijmegen questionnaire HUFA deficiency questionnaire

Reading and writing tests:

DLS etc

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 8-18 years
* Met DSM-IV criteria for a diagnosis of ADHD of any subtype

Exclusion Criteria:

* Autism
* Psychosis
* Bipolar disorder
* Mental retardation
* Uncontrolled seizure disorder
* Hyper- or hypothyroidism
* Significant other medical conditions
* Weight below 20 kg
* Alcohol or drug abuse or the use in the past three months of any psychoactive drugs or Omega 3 preparations

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2004-08; Primary Completion 2006-06 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
ADHD-Rating Scale, Investigator-rated | From 0-3 months
  The scale comprises the 18 DSM-IV items included in the ADHD diagnosis, and each item is assessed on a 0-3 point scale
ADHD-Rating Scale, Investigator-rated | From 3-6 months
  The scale comprises the 18 DSM-IV items included in the ADHD diagnosis, and each item is assessed on a 0-3 point scale

SECONDARY OUTCOMES:
Clinical Global Impression-Severity Scale | From 0-3 months
  Investigator-rated global impression of ADHD symptom severity
Clinical Global Impression-Severity Scale | From 3-6 months
  Investigator-rated global impression of ADHD symptom severity

CONTACTS AND LOCATIONS:
Overall Officials: Mats Johnson, MD, Principal Investigator — Göteborg University

REFERENCES:
- [Derived] Johnson M, Mansson JE, Ostlund S, Fransson G, Areskoug B, Hjalmarsson K, Landgren M, Kadesjo B, Gillberg C. Fatty acids in ADHD: plasma profiles in a placebo-controlled study of Omega 3/6 fatty acids in children and adolescents. Atten Defic Hyperact Disord. 2012 Dec;4(4):199-204. doi: 10.1007/s12402-012-0084-4. Epub 2012 Jul 3. PMID 22753087